CLINICAL TRIAL: NCT06141694
Title: Assessment of Clinical Capabilities of LIBERTY® Endovascular Robotic System's Performance and Safety in Peripheral Vascular Interventions: A Multi-Center, Single Arm, Prospective Trial (ACCESS-PVI)
Brief Title: Assessment of Clin. Capabilities of LIBERTY® Endovascular Robotic System's Performance & Safety in Periph. Vasc. Interv.
Acronym: ACCESS-PVI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Microbot Medical, INC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CLN-001P
Record Dates: First submitted 2023-11-15; First posted 2023-11-21 (Actual); Last update posted 2024-10-17 (Actual); Status verified 2024-10

CONDITIONS: Peripheral Vascular Interventions

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- Endovascular Robotic Navigation (Experimental)
  Interventions: Device: The LIBERTY® Robotic System

INTERVENTIONS:
Device: The LIBERTY® Robotic System — The LIBERTY® Robotic System is intended for use in the remote delivery and manipulation of guidewires and catheters, and remote manipulation of guide catheters, to facilitate navigation to anatomical targets in the peripheral vasculature.
  The LIBERTY® Robotic System is not intended for coronary or neurointerventional procedures.

SUMMARY:
A prospective, multi-center, single-arm, study to evaluate the performance and safety of the LIBERTY® Robotic System in human subjects undergoing Peripheral Vascular Interventions. The study is designed to evaluate the performance and safety of endovascular procedures supported by the LIBERTY® Robotic System. The System is configured to deliver and manipulate third-party commercially available surgical devices that are employed in endovascular transcatheter procedures (guidewires, microcatheters, and guiding catheters).

ELIGIBILITY:
Inclusion Criteria:

1. The subject is age 22-80 years at screening.
2. The subject has been informed of the nature of the study and is willing and able to provide informed consent to participate in the study.
3. The subject has a clinical indication for an elective PVI.
4. The subject is willing and able to comply with all required study procedures.
5. Subject's scheduled procedure is compatible with commercially available peripheral interventional devices that have the following diameter ranges:

   1. Guidewires: 0.014-0.018"
   2. Catheters (Microcatheters): 2-3 Fr
   3. Guide catheter: 4-6 Fr

Exclusion Criteria:

1. Subject is planned to undergo coronary and/or neuro-interventional procedures during study procedure.
2. Subject with vasculature that cannot accommodate the catheter or required accessories according to local routine practice guidelines.
3. Subject with contraindication to endovascular approach to the treatment of peripheral vascular disease, similar or same as contraindications in manual procedures.
4. Target vessel has been previously treated with any type of a bypass conduit.
5. Subject has a contraindication to standard anticoagulation for PVIs.
6. Subject has bleeding or a hypercoagulability disorder.
7. Subject has thrombocytopenia (<50 x103 per µL).
8. Subject has abnormal, clinically relevant lab results resulting in treatment and/or increased risk to the subject.
9. Subject has an elevated serum creatinine (≥2.5 mg/dL or ≥221 mmol/L).
10. Subject has an active infection requiring antibiotic or anti-fungal systemic treatment.
11. Subject has a known allergy to any material used or any component of the devices used that will be in direct contact with subject's tissue.
12. Subject is pregnant or lactating.
13. Subject with any medical, social, or psychological conditions which, in the opinion of the investigator, would prohibit appropriate consent or impair completion of the study protocol or study procedures.
14. Subject who is incapable, per the investigator's discretion, of following-up with the study visit schedule for any reason.
15. Subject is currently participating in an investigational drug or device study or post market registry, or participated in another investigational drug or device study within one month prior to enrollment.

Ages: 22 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2024-07-02 (Actual); Primary Completion 2024-10-10 (Actual); Study Completion 2024-10-15 (Actual)

PRIMARY OUTCOMES:
Effectiveness Endpoint | During navigation portion of the procedure.
  Successful robotic navigation of the guidewire and microcatheter is defined as reaching at least 95% of the predetermined anatomical target locations using the LIBERTY® Robotic System, without switching from a robotic to manual procedure due to difficulty reaching the target site.

SECONDARY OUTCOMES:
Safety Endpoint | Through the three (3) day follow-up visit period.
  Safety of the LIBERTY® Robotic System will be evaluated by the number and rate of Adverse Device Effects (ADEs) reported

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - Baptist Hospital of Miami, Miami, Florida
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Memorial Sloan Kettering Cancer Center, New York, New York

IPD SHARING:
Plan to Share IPD: No